CLINICAL TRIAL: NCT03216759
Title: Effects of Comprehensive Intestinal Protection Strategy on Postoperative Intestinal Complications in Patients Undergoing Laparotomy With General Anesthesia
Brief Title: Effects of Comprehensive Intestinal Protection Strategy on Postoperative Intestinal Complications
Acronym: CIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Kexuan Liu, Director, Head of Anesthesiology, Principal Investigator, Clinical Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIPS
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Intestinal Complications; Laparotomy
Keywords: Comprehensive intestinal protection strategy; Intestinal complications; laparotomy
MeSH Terms: interventions — Ischemic Preconditioning; Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Tourniquet would be tied to left upper limb of Patients who undergoing laparotomy for 30 minutes after the induction of anesthesia,but put no press on it. Other processes are consistent with conventional methods.
- intervention (Experimental): 1. After the anesthesia induction and before surgery,the patient's left upper limb was subjected to ischemic preconditioning.
  2. At the beginning of anesthesia induction, 3 μg / kg / h of dexmedetomidine was infused and adjusted to 0.3 ug / kg / h after 10 min of infusion until 30 minutes before the end of the procedure.
  3. Before the induction of anesthesia, the steel wire epidural catheter was placed in the T8-9 or T10-11 gap.
  Interventions: Procedure: Ischemic preconditioning; Drug: Dexmedetomidine; Procedure: Patient-controlled epidural analgesia

INTERVENTIONS:
Procedure: Ischemic preconditioning — After the anesthesia induction and before surgery,the patient's left upper limb was subjected to ischemic preconditioning then patients received ischemic preconditioning.
  Arms: intervention
Drug: Dexmedetomidine — At the beginning of anesthesia induction, 3 ug/kg/h of dexmedetomidine was infused and adjusted to 0.3 ug/kg/h after 10 min of infusion until 30 minutes before the end of the procedure.
  Arms: intervention
Procedure: Patient-controlled epidural analgesia — Before the induction of anesthesia, the steel wire epidural catheter was placed in the T8-9 or T10-11 gap.The first volume of morphine 2mg + 0.2% ropivacaine + 0.9% saline 6ml, maintenance dose of morphine 18mg + 0.1% ropivacaine + 0.9% saline total 150ml. PCEA work with a continuous background dose of 2 ml/h with a single dose of 2ml/time, load 2ml, locking time 15min.
  Arms: intervention

SUMMARY:
To investigate the morbidity of intestinal injury after open surgery and observe the effect of comprehensive intestinal protection strategy on postoperative intestinal complications in patients undergoing laparotomy with general anesthesia.

DETAILED DESCRIPTION:
Perioperative intestinal injury is one of the common tissues and organs injury in surgical practice. However, there is a lack of effective means of prevention and treatment.The investigators previously found that ischemic preconditioning, IPC, and dexmedetomidine has protective effects on intestinal mucosal injury.

However, the combined effect of various factors has not been clinically validated. To explore the effect of comprehensive intestinal protection strategy on postoperative intestinal complications in patients undergoing laparotomy with general anesthesia,the investigators select the patients undergoing open surgery under general anesthesia as the study subjects and the concentration of intestinal fatty acid binding protein (I-FABP) as well as the incidence of digestive system complications in one week after operation are the main observation indexes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years;
* Elective abdominal surgery under general anesthesia, operation time > 2h;
* ASA Ⅰ ~ Ⅲ;
* Patient informed and consent to accept the test.

Exclusion Criteria:

* persons under the age of 18 or over 70 years old;
* pregnant or lactating women;
* combined with lung, liver, kidney, cardiovascular and hematopoietic system disease and other serious primary disease;
* preoperative Hb <7g / l;
* oral sulfa drugs or nicorandil antihypertensive drugs;
* lower extremity amputees;
* with peripheral vascular disease;
* patients with mental illness or severe neurosis;
* can not express the subjective symptoms;
* nearly 3 months to participate in other drug clinical trials;
* within 3 months of receiving other surgical treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of digestive system complications after operation | 12 hours to one week after surgery
  The incidence of digestive system complications within one week after surgery
The concentration of intestinal fatty acid-binding protein (I-FABP) | 12 h after operation
  The concentration of intestinal fatty acid-binding protein (I-FABP) at 12 h after operation

SECONDARY OUTCOMES:
Postoperative heart and respiratory complications within one week | 12 hours to one week after surgery
  Postoperative heart and respiratory complications within one week

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Xuan Liu, Ph.D, Principal Investigator — Nanfang Hospital, the Southern Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walsh SR, Sadat U, Boyle JR, Tang TY, Lapsley M, Norden AG, Gaunt ME. Remote ischemic preconditioning for renal protection during elective open infrarenal abdominal aortic aneurysm repair: randomized controlled trial. Vasc Endovascular Surg. 2010 Jul;44(5):334-40. doi: 10.1177/1538574410370788. Epub 2010 May 18. PMID 20484066
- [Result] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752